CLINICAL TRIAL: NCT04181125
Title: "Evaluation of Postural Control in Children With Increased Femoral Anteversion"
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Lecturer in Department of Physiotheray and Rehabilitation, Bezmialem Vakif University, Bezmialem Vakif University
Other Study IDs: DT-01
Record Dates: First submitted 2019-11-22; First posted 2019-11-29 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Femoral Anteversion; Gait Disorders in Children; Postural Control; Postural Stability; Balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- Children with increased femoral anteversion: After the demographic information, developmental history and gait information were recorded with the Evaluation Form, clinical evaluation was performed; bilateral lower extremity range of motion, flexibility, leg length measurement, and muscle strength measurement and muscular endurance tests (abdominal, back and lower extremity) will be performed. For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) and the Biodex Balance System for computerized evaluation will be used.
  Interventions: Other: Biodex Balance System; Other: Balance Error Scoring System (BESS)
- Healthy children: After the demographic information, developmental history and gait information were recorded with the Evaluation Form, clinical evaluation was performed; bilateral lower extremity range of motion, flexibility, leg length measurement, and muscle strength measurement and muscular endurance tests (abdominal, back and lower extremity) will be performed. For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) and the Biodex Balance System for computerized evaluation will be used.
  Interventions: Other: Biodex Balance System; Other: Balance Error Scoring System (BESS)

INTERVENTIONS:
Other: Biodex Balance System — For the computerized evaluation of postural control, Biodex Balance System will be used.
Other: Balance Error Scoring System (BESS) — For the clinical evaluation of postural control, the Modified Balance Error Scoring System (BESS) will be used.

SUMMARY:
The relationship between increased femoral anteversion and postural control in healthy children has not been studied in the current literature. To our knowledge there is no study to evaluate postural control in children with increased femoral anteversion by computerized posturography. We aimed to evaluate postural control in children with increased femoral anteversion using computerized dynamic posturography (Biodex Balance System).

DETAILED DESCRIPTION:
Femoral anteversion is defined as the angle formed by the femoral condyles plane (bicondylar plane) and a plane passing through the center of the neck and femoral head. Toe-in-gait pattern may be due to foot deformity (metatarsus adductus) and / or abnormal transverse alignment of long bones (tibial torsion and / or increased femoral anteversion). Transverse plane deviations are frequently seen in infants and usually improve with typical physiological growth mechanisms. Persistent transverse plan disorder may lead to gait dysfunction. The most important function of the posture is to maintain the balance during the initiation and continuation of the movement. Postural control regulates maintaining the balance and keeping the center of gravity within the body's stability limits. It includes resistance to gravity forces and mechanical support during movement. Postural control is an integral part of achieving targeted action. To our knowledge the relationship between increased femoral anteversion and postural control in healthy children has not been studied in the current literature. Postural control in children with increased femoral anteversion was evaluated by computerized posturography. In this study, we aimed to evaluate postural control in children with increased femoral anteversion using computerized dynamic posturography (Biodex Balance System).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as bilateral increased femoral anteversion
* No history of neurological, psychiatric diseases
* Lack of intellectual disability to prevent evaluation and treatment participation
* No participation in any physiotherapy program in the last six months
* Written permission from the parents for participate in the study

Exclusion Criteria:

* History of surgery or BoNT-A for lower extremities
* Leg length discrepancy

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 16 children with bilateral increased femoral anteversion aged 6-15 years followed by Bezmialem Vakıf University Department of Orthopedics and Traumatology.
  16 healthy volunteers aged 6-15 years will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Postural control-postural stability | 1 day
  Computerized test of postural stability with Biodex Balance System
Postural control-limits of stability | 1 day
  Computerized test of limits of stability with Biodex Balance System
Postural control-sensory integration | 1 day
  Computerized test of sensory integration with Biodex Balance System
Balance Error Scorring System-BESS | 1 day
  Clinical evaluation of postural control

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Nilgun Gurses, Prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)